CLINICAL TRIAL: NCT02512315
Title: 4 Cycles Of Neoadjuvant Chemotherapy Plus Concurrent Chemoradiation Versus Concurrent Chemoradiation Alone In Patients With Stage N2-3 Nasopharyngeal Carcinoma: A Phase 3 Multicenter Randomised Controlled Trial
Brief Title: A Trial On 4 Cycles Of Neoadjuvant Chemotherapy Plus Concurrent Chemoradiation In N2-3 Nasopharyngeal Carcinoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yuan-hong Gao, Deputy Director of Department of Radiation Oncology, Sun Yat-sen University Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NACT4-NPC-5010
Record Dates: First submitted 2015-07-24; First posted 2015-07-30 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Nasopharyngeal carcinoma; Neoadjuvant chemotherapy; Concurrent chemoradiation; Distant metastasis; Survival
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CCRT group (Group A) (Active Comparator): Patients who are allocated into in this group will be treated with concurrent chemoradiation (CCRT).
  Interventions: Radiation: Concurrent chemoradiation (CCRT)
- NACT-CCRT group (Group B) (Experimental): Patients who are allocated into in this group will be treated with 4 cycles of neoadjuvant chemotherapy (NACT, docetaxel plus cisplatin) followed by CCRT.
  Interventions: Drug: Docetaxel (DOC); Drug: Cisplatin (DDP); Radiation: Concurrent chemoradiation (CCRT)

INTERVENTIONS:
Drug: Docetaxel (DOC) — Neoadjuvant chemotherapy (NACT) is administrated every 3 weeks with the regimen comprised of docetaxel plus cisplatin. A total of 4 cycles of NACT is applied. Docetaxel is given at a dose of 75mg/m2 on the first day of every cycle.
  Other Names: Docetaxel Injection
  Arms: NACT-CCRT group (Group B)
Drug: Cisplatin (DDP) — Neoadjuvant chemotherapy (NACT) is administrated every 3 weeks with the regimen comprised of docetaxel plus cisplatin. A total of 4 cycles of NACT is applied. Cisplatin is given at a dose of 75mg/m2 on the first day of every cycle.
  Other Names: Cisplatin Injection
  Arms: NACT-CCRT group (Group B)
Radiation: Concurrent chemoradiation (CCRT) — The technology of radiotherapy is intensity-modulated radiation therapy (IMRT). A total dose of 66-72Gy is given to gross tumor of nasopharynx (GTVnx), 60-70Gy to positive neck lymph nodes (GTVnd), 60Gy to high-risk region (CTV1), and 50-54Gy to prophylactic irradiation region (CTV2).
  The regimen of concurrent chemotherapy is single-agent cisplatin 40mg/m2 weekly.

SUMMARY:
The standard treatment strategy of locally advanced nasopharyngeal carcinoma (NPC) nowadays is concurrent chemoradiation (CCRT) based on intensity-modulated radiation therapy (IMRT). However, distant metastasis remains the major cause of treatment failure, especially in patients with T1-4N2-3M0 diseases (N2-3 NPC). The investigators inferred that it was more appropriate to consider N2-3 NPC as a systemic disease instead of a local disease. NACT of sufficient intensity such as 4 cycles might be effective enough for control of the pre-existing micrometastases. Therefore, the objective of this phase 3 multicenter randomized controlled trial is to make a comparison between NACT of 4 cycles plus CCRT based on IMRT and CCRT alone in N2-3 NPC on distant metastasis, survival and adverse reaction.

DETAILED DESCRIPTION:
The standard treatment strategy of locally advanced nasopharyngeal carcinoma (NPC) nowadays is concurrent chemoradiation (CCRT), which is based on intensity-modulated radiation therapy (IMRT) and achieves a satisfactory local-regional control and a 5-year overall survival (OS) of 83.0%. However, distant metastasis remains the major cause of treatment failure, especially in patients with T1-4N2-3M0 diseases (N2-3 NPC). The distant metastasis reaches 35-48% after CCRT alone.

To decrease distant metastasis of locally advanced NPC so as to improve survival, approaches on modifying timing of chemotherapy have been made to mainly 2 types: one was CCRT plus adjuvant chemotherapy (ACT), the other was neoadjuvant chemotherapy (NACT) plus CCRT. It was proved that CCRT plus ACT could not improve survival of locally advanced NPC further. Some clinical trials indicated that locally advanced NPC patients with 2-3 cycles of NACT plus CCRT had a better survival than those with CCRT alone though the roles of NACT remain controversial.

It is known that N stage is by far the most significant predicting factor of metastasis risk for NPC. N2-3 NPC was also proved to have a quite great risk of distant failure. 51.4% of distant metastases happened within 1 year after CCRT. The investigators inferred that subclinical micrometastases were already present before treatment starting. Hence, it was more appropriate to consider N2-3 NPC as a systemic disease instead of a local disease. NACT of sufficient intensity such as 4 cycles might be effective enough for control of the pre-existing micrometastases.

Therefore, this phase 3 multicenter randomized controlled trial is conducted to enroll 144 patients with N2-3 NPC. After stratification by N stage, the patients will be allocated into 2 treatment groups randomly at a ratio of 1:1 and applied with different treatment strategies to make a comparison between NACT of 4 cycles plus CCRT based on IMRT and CCRT alone in N2-3 NPC on distant metastasis, survival and adverse reaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pathological diagnosis of nasopharyngeal carcinoma
* Union Internationale Contre le Cancer/American Joint Cancer Committee (UICC/AJCC) 2010 Stage T1-4 N2-3 M0 through magnetic resonance imaging of head and neck, whole-body bone scan and thoracoabdominal computed tomography
* Male or female with age no older than 70 years old
* Karnofsky Performance Scores ≥ 80
* Expected survival ≥ 3 months

Exclusion Criteria:

* Patients with distant metastasis before or during radiotherapy
* Severe dysfunction of heart, lung, liver, kidney or hematopoietic system
* Severe neurological, mental or endocrine diseases
* History of other malignancies
* Prior chemotherapy, radiotherapy or application of monoclonal antibodies
* Patients participated in clinical trials of other drugs within last 3 months
* Pregnant or lactating women
* Those who are considered by the researchers unsuitable to participate

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
5-year overall survival (5y-OS) | 5 years after the date of pathologic diagnosis
  Percentage of patients in a treatment group who are alive for a 5-year period of follow-up after the date of pathologic diagnosis
5-year distant-metastasis-free survival (5y-MFS) | 5 years after the date of pathologic diagnosis
  Percentage of patients in a treatment group who are alive without distant metastasis for a 5-year period of follow-up after the date of pathologic diagnosis

SECONDARY OUTCOMES:
5-year local-relapse-free survival (5y-RFS) | 5 years after the date of pathologic diagnosis
  Percentage of patients in a treatment group who are alive without local recurrence for a 5-year period of follow-up after the date of pathologic diagnosis
5-year disease-free survival (5y-DFS) | 5 years after the date of pathologic diagnosis
  Percentage of patients in a treatment group who are alive without disease-related events (local recurrence, distant metastasis) for a 5-year period of follow-up after the date of pathologic diagnosis
Incidence of grade 3/4 adverse event | Once a week during therapy, up to 7 weeks (Group A) or 19 weeks (Group B)
  Incidence of patients in a treatment group who manifest a specific adverse event (such as myelosuppression) of grade 3/4. Incidence is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 4.0 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-hong Gao, M.D, Principal Investigator — Sun Yat-sen University
Locations (4):
- China (4):
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong

REFERENCES:
- [Background] Moss WT. Therapeutic radiology, 2nd ed. St Louis, MO: Mosby; 1965: 142-180.
- [Background] Guigay J, Temam S, Bourhis J, Pignon JP, Armand JP. Nasopharyngeal carcinoma and therapeutic management: the place of chemotherapy. Ann Oncol. 2006 Sep;17 Suppl 10:x304-7. doi: 10.1093/annonc/mdl278. No abstract available. PMID 17018743
- [Background] Al-Sarraf M, LeBlanc M, Giri PG, Fu KK, Cooper J, Vuong T, Forastiere AA, Adams G, Sakr WA, Schuller DE, Ensley JF. Chemoradiotherapy versus radiotherapy in patients with advanced nasopharyngeal cancer: phase III randomized Intergroup study 0099. J Clin Oncol. 1998 Apr;16(4):1310-7. doi: 10.1200/JCO.1998.16.4.1310. PMID 9552031
- [Background] Lin JC, Jan JS, Hsu CY, Liang WM, Jiang RS, Wang WY. Phase III study of concurrent chemoradiotherapy versus radiotherapy alone for advanced nasopharyngeal carcinoma: positive effect on overall and progression-free survival. J Clin Oncol. 2003 Feb 15;21(4):631-7. doi: 10.1200/JCO.2003.06.158. PMID 12586799
- [Background] Wee J, Tan EH, Tai BC, Wong HB, Leong SS, Tan T, Chua ET, Yang E, Lee KM, Fong KW, Tan HS, Lee KS, Loong S, Sethi V, Chua EJ, Machin D. Randomized trial of radiotherapy versus concurrent chemoradiotherapy followed by adjuvant chemotherapy in patients with American Joint Committee on Cancer/International Union against cancer stage III and IV nasopharyngeal cancer of the endemic variety. J Clin Oncol. 2005 Sep 20;23(27):6730-8. doi: 10.1200/JCO.2005.16.790. PMID 16170180
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] J. Y. Hsiang, K. Liu, S. Iganej, et al. Concurrent chemoradiation with and without adjuvant chemotherapy in advanced stage nasopharyngeal carcinoma: A retrospective analysis. J Clin Oncol. 2004, 22(Supp 114): 5619.
- [Background] Pignon JP, le Maitre A, Maillard E, Bourhis J; MACH-NC Collaborative Group. Meta-analysis of chemotherapy in head and neck cancer (MACH-NC): an update on 93 randomised trials and 17,346 patients. Radiother Oncol. 2009 Jul;92(1):4-14. doi: 10.1016/j.radonc.2009.04.014. Epub 2009 May 14. PMID 19446902
- [Background] Tan T, Lim WT, Fong KW, Cheah SL, Soong YL, Ang MK, Ng QS, Tan D, Ong WS, Tan SH, Yip C, Quah D, Soo KC, Wee J. Concurrent chemo-radiation with or without induction gemcitabine, Carboplatin, and Paclitaxel: a randomized, phase 2/3 trial in locally advanced nasopharyngeal carcinoma. Int J Radiat Oncol Biol Phys. 2015 Apr 1;91(5):952-60. doi: 10.1016/j.ijrobp.2015.01.002. PMID 25832687
- [Background] Hui EP, Ma BB, Leung SF, King AD, Mo F, Kam MK, Yu BK, Chiu SK, Kwan WH, Ho R, Chan I, Ahuja AT, Zee BC, Chan AT. Randomized phase II trial of concurrent cisplatin-radiotherapy with or without neoadjuvant docetaxel and cisplatin in advanced nasopharyngeal carcinoma. J Clin Oncol. 2009 Jan 10;27(2):242-9. doi: 10.1200/JCO.2008.18.1545. Epub 2008 Dec 8. PMID 19064973
- [Background] Loong HH, Ma BB, Leung SF, Mo F, Hui EP, Kam MK, Chan SL, Yu BK, Chan AT. Prognostic significance of the total dose of cisplatin administered during concurrent chemoradiotherapy in patients with locoregionally advanced nasopharyngeal carcinoma. Radiother Oncol. 2012 Sep;104(3):300-4. doi: 10.1016/j.radonc.2011.12.022. Epub 2012 Jan 31. PMID 22300609
- [Background] Honkoop AH, Luykx-de Bakker SA, Hoekman K, Meyer S, Meyer OW, van Groeningen CJ, van Diest PJ, Boven E, van der Wall E, Giaccone G, Wagstaff J, Pinedo HM. Prolonged neoadjuvant chemotherapy with GM-CSF in locally advanced breast cancer. Oncologist. 1999;4(2):106-11. PMID 10337380
- [Background] da Costa Miranda V, de Souza Fede AB, Dos Anjos CH, da Silva JR, Sanchez FB, da Silva Bessa LR, de Paula Carvalho J, Filho EA, de Freitas D, Del Pilar Estevez Diz M. Neoadjuvant chemotherapy with six cycles of carboplatin and paclitaxel in advanced ovarian cancer patients unsuitable for primary surgery: Safety and effectiveness. Gynecol Oncol. 2014 Feb;132(2):287-91. doi: 10.1016/j.ygyno.2013.12.002. Epub 2013 Dec 9. PMID 24333355
- [Background] Sun XM, Huang Y, Chen CY, et al. Long-term outcomes of patients with advanced N-stage nasopharyngeal carcinoma treated by intensity-modulated radiotherapy alone or with chemotherapy. Chinese Journal of Radiation Oncology. 2013, 22(3): 225-229.
- [Background] Ghossein RA, Bhattacharya S, Rosai J. Molecular detection of micrometastases and circulating tumor cells in solid tumors. Clin Cancer Res. 1999 Aug;5(8):1950-60. PMID 10473071
- [Background] Lee AW, Au JS, Teo PM, Leung TW, Chua DT, Sze WM, Zee BC, Law SC, Leung SF, Tung SY, Kwong DL, Lau WH. Staging of nasopharyngeal carcinoma: suggestions for improving the current UICC/AJCC Staging System. Clin Oncol (R Coll Radiol). 2004 Jun;16(4):269-76. doi: 10.1016/j.clon.2004.01.008. PMID 15214651
- [Background] Gao J, Tao YL, Li G, Yi W, Xia YF. Involvement of difference in decrease of hemoglobin level in poor prognosis of Stage I and II nasopharyngeal carcinoma: implication in outcome of radiotherapy. Int J Radiat Oncol Biol Phys. 2012 Mar 15;82(4):1471-8. doi: 10.1016/j.ijrobp.2011.05.009. Epub 2011 Jun 25. PMID 21708429
- [Derived] Xie WH, Xiao WW, Chang H, Xu MJ, Hu YH, Zhou TC, Zhong Q, Chen CY, Lu LX, Wang QX, Zhu YJ, Yang J, Shi XY, Kang HL, Wei JW, Huang R, Peng HH, Yuan Y, Wu SH, Jiang XH, Liu YJ, Wen BX, Gao YH. Four cycles of docetaxel plus cisplatin as neoadjuvant chemotherapy followed by concurrent chemoradiotherapy in stage N2-3 nasopharyngeal carcinoma: phase 3 multicentre randomised controlled trial. BMJ. 2025 Apr 15;389:e081557. doi: 10.1136/bmj-2024-081557. PMID 40233976